CLINICAL TRIAL: NCT02705911
Title: Isometric Handgrip Exercise: a New Non-pharmacological Tool in the Management of High Blood Pressure?
Brief Title: TeleRehabilitation in Hypertension
Acronym: TRiHYP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Véronique Cornelissen, PhD, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1502214N
Record Dates: First submitted 2016-03-03; First posted 2016-03-11 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Hypertension; Pre-hypertension; Healthy
MeSH Terms: conditions — Hypertension; Prehypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Isometric Handgrip training (Experimental): Participants are asked to perform daily 4 x 2 minute contractions with alternating hands , separated with 1 minute rest period using a ZonaHealth device;
  Interventions: Other: Isometric handgrip exercise
- Aerobic endurance training (Active Comparator): Participants are asked to perform at least 150 minutes extra of moderate aerobic exercise per week
  Interventions: Other: Aerobic endurance training
- Control (No Intervention): Participants are asked to continue with their daily routine and not to perform extra exercise.

INTERVENTIONS:
Other: Isometric handgrip exercise — Participants have to perform 4 x 2 minute contractions with alternating hands, separated with 1 minute rest period using a ZonaHealth device;
  Arms: Isometric Handgrip training
Other: Aerobic endurance training — To perform 150 minutes extra/week at moderate aerobic intensity
  Arms: Aerobic endurance training

SUMMARY:
The purpose of this RCT which will be performed in 60 healthy adults is I. To assess the training effects of 8 weeks of isometric handgrip exercise on BP; and to test whether it yields at least similar effects on BP compared to current exercise recommendations.

II. To assess whether isometric handgrip training yields larger BP reductions beyond the supervised training period at 6 months of follow-up.

III. To determine whether changes in BP following acute exercise and chronic training can be explained by changes in important physiological mechanisms known to mediate or to be associated with BP?

ELIGIBILITY:
Inclusion Criteria:

* not physically active (< 3 hours of moderate to high levels of PA/week) low cardiovascular risk according to current guidelines (Mancia et al J Hypertens 2013) will be recruited through advertisements. The latter is defined as:
* >115 mmHg < systolic BP < 139 mmHg and/or 75 mmHg< diastolic BP<90mmHg in the presence of 0 to a maximum of three other cardiovascular risk factors, excluding diabetes Or
* 139 mmHg < systolic BP < 160 mmHg and/or 90 mmHg<DBP< 100 mmHg in the absence of other cardiovascular risk factors

Exclusion Criteria:

* current smoker
* pregnancy
* presence of other cardiovascular disease, pulmonary disease or metabolic disease
* inability to perform a standard exercise program due to mental/physical disability.
* use of antihypertensive drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
change in office blood pressure at 8 weeks of follow-up | 8 weeks - 6 months

SECONDARY OUTCOMES:
change in exercise tolerance (peakVO2 in ml/min/kg) at 8 weeks of follow-up | 8 weeks - 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium